CLINICAL TRIAL: NCT06849752
Title: EAGLE-HF is Part of a Multinational Group of Studies Titled; Screening for Early Heart Failure Diagnosis and Management in Primary Care or at Home Using Natriuretic Peptides and Echocardiography
Brief Title: Early Assessment and Initiation of GuideLine-Directed Evidence-Based Management-HF
Acronym: EAGLE-HF
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: University of Glasgow (Other); Roche Diagnostics GmbH (Industry); EchoNous Inc. (Industry)
Responsible Party: Principal Investigator, Nancy M. Albert, Ph.D., Associate Chief Nursing Officer-Research and Innovation; Senior Nurse Scientist, The Cleveland Clinic
Other Study IDs: 23-423
Record Dates: First submitted 2024-04-20; First posted 2025-02-27 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure; Socioeconomic Adversity
Keywords: medication prescribing; NTproBNP; Provider type; Social determinants of health
MeSH Terms: conditions — Heart Failure; Financial Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — NTproBNP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Test used to diagnose heart failure (NTproBNP) group: Will have a NTproBNP blood test completed at baseline if in the ACTIVE SYMPHONY arm. Baseline NTproBNP test results will be used to assess EAGLE-HF outcomes regarding optimal test cut points for (a) heart failure diagnosis; (b) based on each of the 6 social determinants of health and totla number of social determinants of health; (c) based on risk factors and (d) based on medical comorbidities.
- Participants with heart failure diagnosis: Medication prescribing patterns in the first 6 months after HFrEF diagnosis will be assessed for association with (a) social vulnerability index, (b) distressed community index, (c) physician practice type (Internal Medicine, Cardiology, HF Cardiology or other provider); and (d) medical provider type (physician, advance practice provider [APP] or PharmD)
- Social determinants of health: All participants will be assessed to determine if 6 factors: race, social vulnerability index (SVI), marital status, comfort living on income, distressed community index (DCI) and insurance type are associated with future assessment of HF via biomarkers (troponin or NT-proBNP) and/or echocardiography over the 5 year assessment period

SUMMARY:
EAGLE-HF (Early Assessment and initiation of GuideLine-directed Evidence-based management-HF) is a prospective single site study of a multinational, unblinded, randomized-controlled, longitudinal trial called SYMPHONY. Primary, secondary and exploratory outcomes that are part of SYMPHONY are not described herein as they replicate SYMPHONY outcomes. Data associated with SYMPHONY outcomes will be sent to the SYMPHONY coordinating center. In EAGLE-HF, site investigators will examine if a new-onset heart failure (HF) diagnosis are asscoiated with social determinants of health (6 factors), social vulnerability index and distressed community indices. In addition, for patients diagnosed with HFrEF, prescribing patterns (use of and dose of) core HF medications will be assessed for association with physician practice type and medical provider type. Finally, (among participants in the SYMPHONY Active arm, an optimal NTproBNP cut-point will be assessed for diagnosis of HF based on social determinants of health, social vulnerability index, distressed community index, HF risk factors and medical comorbidities.

DETAILED DESCRIPTION:
EAGLE-HF (Early Assessment and initiation of GuideLine-directed Evidence-based management-HF) is a prospective single site observational study of a multinational, unblinded, randomized-controlled, longitudinal trial called SYMPHONY. Primary, secondary and exploratory outcomes that are part of SYMPHONY are not described herein as they replicate SYMPHONY outcomes (available in clinicaltrials.gov). EAGLE-HF is a prospective observational design involving SYMPHONY participants. In EAGLE-HF, patients from SYMPHONY will make up 3 cohorts: all SYMPHONY participants from our site (n=1000), those who had a NT-proBNP test completed (n=500), and those diagnosed with heart failure (unknown, but approximately =50+). EAGLE-HF specific endpoints include examining if social determinants of health (6 factors), social vulnerability index component and overall scores and distressed community index component and overall scores are associated with new onset heart failure. Among patients with NTproBNP data, optimal cut-points for diagnosis of HF will be assessed, including if optimal cut-points are based on social determinants of health, social vulnerability score, distressed community score, risk factors for developing HF and medical comorbidities. Finally, in SYMPHONY participants who are diagnosed with HFrEF within 6 months of enrollment, medication prescribing patterns (use and dose of 4 classes of core HFrEF medications) will be examined, the site investigators will assess if medication prescribing patterns are based on physician practice type and medical provider type.

ELIGIBILITY:
Inclusion Criteria are patients enrolled in SYMPHONY as described below:

* ≥40 years old at enrollment
* Willing to sign informed consent
* Specific Activity Scale results that match a NYHA-FC score II-IV
* Has a minimum of 2 documented risk factors for heart failure:
* Established cardiovascular disease (e.g. persistent or permanent atrial fibrillation, myocardial infarction/ coronary artery disease [coronary artery bypass grafting, percutaneous coronary intervention or documented stenosis or an epicardial coronary artery (50% LMS, >70% LAD/Cx/RCA], or valvular heart disease)
* An established diagnosis of diabetes (type I or II)
* Persistent or permanent atrial fibrillation (NOT paroxysmal atrial fibrillation)
* Previous ischemic or embolic stroke
* Peripheral arterial disease (previous surgical or percutaneous revascularisation or a documented stenosis > 50% of a major peripheral arterial vessel).
* Chronic kidney disease (defined as an estimated glomerular filtration rate <60 mL/min/1.73m2 or eGFR 60-90 mL/min/1.73m2 and UACR > 300 mg/g)
* Loop diuretic use for > 30 days (reported at any time in the 12 months prior to consent)
* Chronic obstructive pulmonary disease (COPD; evidenced by one of the following; PFTs showing airway obstruction, diagnosis by respiratory physician, CT scan reporting presence of emphysema or treatment with national guideline advocated COPD therapy).

Exclusion Criteria:

* Inability to give informed consent; e.g., due to significant cognitive impairment, low English proficiency, inability to read, and/or inability to understand consent content or explanations provided by investigators
* Previous diagnosis of HF (with any ejection fraction and due to any cause)
* Receiving renal replacement therapy
* Inability to travel to Cleveland Clinic for biomarker or handheld point-of-care echo with AI (receiving hospice or skilled nursing facility care).
* Anyone who, in the investigators' opinion, is not suitable to participate in the trial for other reasons e.g. a diagnosis which may compromise survival over the study period; female with a history of left breast mastectomy and breast reconstruction (inability to use AI echocardiogram) or history of only 1 visit to Cleveland Clinic for medical care in any service or with any provider (reflects a lack of using Cleveland Clinic for routine medical care)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among adutls enrolled in SYMPHONY (Glasgow, UK), the EAGLE-HF component will use available data; specifically, NTproBNP, HFrEF diagnosis, 4 classes of HF medications use in first 6 months after diagnosis and race, plus data collected locally for EAGLE-HF on social vulnerability index (SVI), marital status, comfort living on income, distressed community index (DCI), insurance type; physician practice type and medical provider type. to determine if variables are associated with EAGLE-HF outcomes
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
New onset HF based on race | 5 years
  Race (a categorical variable) may be reduced to white vs. all other if other categories have too low a sample size. New-onset heart failure is based on electronic health record documentation of elevated NTproBNP and/or echocardiography results + patient symptoms.
New onset HF based on social vulnerability index | 5 years
  SVI (national data based on zip code) Scores range from 0 to 1, with lower scores equating to less social vulnerability. Note: scores may be categorized into SVI factors are socioeconomic status, household characteristics, racial and ethnic minority status, and housing type and transportation that has 4 categories from low vulnerability to high vulnerability). New onset heart failure is based on electronic health record documentation of elevated NTproBNP and/or echocardiography results + patient symptoms.
New onset HF based on marital status | 5 years
  Marital status (a categorical variable that may be reduced to married vs. not married) if other categories have too low of a sample size. New onset heart failure is based on electronic health record documentation of elevated NTproBNP and/or echocardiography results + patient symptoms.
New onset HF based on patients comfort living on income | 5 years
  Comfort living on income is a single patient reported outcome measure with 3 response options: less than comfortable, comfortable, more than comfortable.New onset heart failure is based on electronic health record documentation of elevated NTproBNP and/or echocardiography results + patient symptoms.
New onset HF based on distressed community index (DCI) | 5 years
  DCI (national database information based on zip code) with 7 categories of data based on home location. Scores are from 0-100 with higher scores equating to a more distressed community. Results can be categorized on 5 levels from distressed to prosperous. New onset heart failure is based on electronic health record documentation of elevated NTproBNP and/or echocardiography results + patient symptoms.
New onset HF based on healthcare insurance type | 5 years
  Insurance type (categorical variable from the hospital billing database that includes government insurance, private insurance, health maintenance organization programs and self-pay), that may be reduced to government vs. other insurance vs. self-pay. New onset heart failure is based on electronic health record documentation of elevated NTproBNP and/or echocardiography results + patient symptoms.
New onset HF based on all 6 social determinants that may affect health | 5 years
  Social determinants of health are defined by results of 6 variables (race, SVI, marital status, comfort living on income, DCI, and insurance type). Each of the 6 variables will receive a score reflecting low, medium or high probability of better health and the combined score will be assessed for association with new onset heart failure over 5 year period (yes/no).

SECONDARY OUTCOMES:
Use of HFrEF core medication classes based on distressed community index (DCI) | 6 months post HFrEF diagnosis
  DCI score (0-100) comes from a national database that uses zip code to determine community distress (previously described). HFrEF medication "use" score is based on prescription of core 4 classes of medications per the electronic health record: 1) renin-angiotensin system inhibitors (RASi) or hydralazine/nitrate if severe chronic kidney disease or other contraindication, 2) evidenced-based beta blockers (eBB) or ivabradine if beta blockers are contraindicated), 3) mineralocorticoid receptor blocker (MRA), and 4) sodium-glucose co-transporter inhibitor (SGLTi); scoring is based on drug class- 1 to 4.
Dose of HFrEF core medication classes based on distressed community index (DCI) | 6 months post HFrEF diagnosis
  DCI score (0-100) comes from a national database that uses zip code to determine community distress (previously described). HFrEF medication "dose" score is based on prescription dose of core 4 classes of medications per the electronic health record: 1) RASi or hydralazine/nitrate if severe chronic kidney disease or other contraindication, 2) eBB or ivabradine if beta blockers are contraindicated), 3) MRA, and 4) SGLTi; scoring has 4 categories: not used, < 50% target dose, 50-100% target dose and > 100% target dose per national HFrEF guidelines
Use of HFrEF core medication classes based on social vulnerability index (SVI) | 6 months post HFrEF diagnosis
  SVI score (0-1) comes from a national database that uses zip code to determine social vulnerability (previously described). HFrEF medication "use" score is based on prescription of core 4 classes of medications per the electronic health record: 1) RASi or hydralazine/nitrate if severe chronic kidney disease or other contraindication, 2) eBB or ivabradine if beta blockers are contraindicated, 3) MRA, and 4) SGLTi; scoring is based on drug class- 1 to 4.
Dose of HFrEF core medication classes based on social vulnerability index (SVI) | 6 months post HFrEF diagnosis
  SVI score (0-1) comes from a national database that uses zip code to determine social vulnerability (previously described). DCI score (0-100) comes from a national database that uses zip code to determine community distress (previously described). HFrEF medication "dose" score is based on prescription dose of core 4 classes of medications per the electronic health record: 1) RASi or hydralazine/nitrate if severe chronic kidney disease or other contraindication, 2) eBB or ivabradine if beta blockers are contraindicated), 3) MRA, and 4) SGLTi; scoring has 4 categories: not used, < 50% target dose, 50-100% target dose and > 100% target dose per national HFrEF guidelines.
Use of HFrEF core medication classes based on medical provider type | 6 months post HFrEF diagnosis
  Medical provider type refers to prescribers of HF medications- 3 categories 1) physician; 2) advanced practice provider (nurse or physician assistant); 3) pharmacist (PharmD). The medication prescribing patterns were previously described as prescription of up to 4 classes of heart failure medications: 1) RASI; 2) eBB; 3) MRA; 4) SGLTi.
Dose of HFrEF core medication classes based on medical provider type | 6 months post HFrEF diagnosis
  Medical provider type refers to prescribers of HF medications- 3 categories 1) physician; 2) advanced practice provider (nurse or physician assistant); 3) pharmacist (PharmD). HFrEF medication "dose" score is based on prescription dose of core 4 classes of medications per the electronic health record: 1) RASi or hydralazine/nitrate if severe chronic kidney disease or other contraindication, 2) eBB or ivabradine if beta blockers are contraindicated), 3) MRA, and 4) SGLTi; scoring has 4 categories: not used, < 50% target dose, 50-100% target dose and > 100% target dose per national HFrEF guidelines.
Use of HFrEF core medication classes based on physician practice type | 6 months post HFrEF diagnosis
  Physician practice type is defined as 1 of 4 categories of primary provider type who manage patients with HFrEF: 1) internal medicine/family practice; 2) cardiology; 3) heart failure specialty cardiology; and 4) other provider. HFrEF medication "use" score is based on prescription of core 4 classes of medications per the electronic health record: 1) RASi or hydralazine/nitrate if severe chronic kidney disease or other contraindication, 2) eBB or ivabradine if beta blockers are contraindicated, 3) MRA, and 4) SGLTi; scoring is based on drug class- 1 to 4.
Dose of HFrEF core medication classes based on physician practice type | 6 months post HFrEF diagnosis
  Physician practice type is defined as 1 of 4 categories of primary provider type who manage patients with HFrEF: 1) internal medicine/family practice; 2) cardiology; 3) heart failure specialty cardiology; and 4) other provider. HFrEF medication "dose" score is based on prescription dose of core 4 classes of medications per the electronic health record: 1) RASi or hydralazine/nitrate if severe chronic kidney disease or other contraindication, 2) eBB or ivabradine if beta blockers are contraindicated), 3) MRA, and 4) SGLTi; scoring has 4 categories: not used, < 50% target dose, 50-100% target dose and > 100% target dose per national HFrEF guidelines.

OTHER OUTCOMES:
Optimal cut-point of NTproBNP for diagnosis of HF in primary care patients meeting study inclusion criteria | Baseline
  In adults who meet inclusion/exclusion criteria for EAGLE-HF and are randomized to the active arm group, NTproBNP mean (standard deviation) values of those who are diagnosed with HF vs. no HF. In those who meet HF criteria (as previously described), cutoff scores may be generated for HFrEF, HFmrEF and HFpEF.
Optimal cut-point of NTproBNP for diagnosis of HF in primary care patients based on social determinants of health (6 factors) | Baseline
  In adults who meet inclusion/exclusion criteria for EAGLE-HF and are randomized to the active arm group, NTproBNP mean (standard deviation) values of those who are diagnosed with HF vs. no HF based on the 6 factors that make up social determinants of health score. Cut-point scores by social determinants of health may be generated for HFrEF, HFmrEF and HFpEF.
Optimal cut-off point of NTproBNP for diagnosis of heart failure in primary care patients based on the number of risk factors for study inclusion (2 to 8) | Baseline
  In adults who are randomized to the active arm group of EAGLE-HF, assess NTproBNP mean (standard deviation) values of those who are diagnosed with HF vs. no HF based on the 8 risk factors for HF development (all patients will have 2 factors and can have up to 8 factors). Cut-point scores by the number of risk factors may be generated for HFrEF, HFmrEF and HFpEF.
Optimal cut-off point of NTproBNP for diagnosis of heart failure in primary care patients based on the 2 most common risk factors for study inclusion | Baseline
  In adults who are randomized to the active arm group of EAGLE-HF, assess NTproBNP mean (standard deviation) values of those who are diagnosed with HF vs. no HF based on the 2 most common risk factors for HF development. Cut-point scores by the 2 most common risk factors may be generated for HFrEF, HFmrEF and HFpEF.
Optimal cut-off point of NTproBNP for diagnosis of heart failure based on medical comorbidity score | Baseline
  In adults who are randomized to the active arm group of EAGLE-HF, assess NTproBNP mean (standard deviation) values of those who develop HF vs. no HF will be compared based on Charlson Co-morbidity Index (CCI) that includes 12 common co-morbid conditions that increase the risk of future morbidity and mortality. A statistician will calculate the CCI score and assess NTproBNP levels based on different CCI categories.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Albert, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Non-EAGLE-HF specific data that is part of SYMPHONY will be deidentified, placed in REDCap, saved as an excel file and will be sent to the SYMPHONY coordinating center every 3 months until all patients are enrolled and 6 month outcomes are completed. After that time, data will be sent at 1, 2 and 5 years post baseline.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 3 months after enrollment and initial visit completion